CLINICAL TRIAL: NCT02825329
Title: Evaluating the Use of Polymyxin B Hemoperfusion in a Prospective Non-controlled Trial in Adults
Brief Title: Open-label Evaluation of Polymyxin B Hemoperfusion for Septic Shock
Acronym: EUPHORIA
Status: Temporarily not available | Type: Expanded Access
Sponsor: Spectral Diagnostics (US) Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SDI-PMX-NA002
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Septic Shock; Endotoxemia
MeSH Terms: conditions — Shock, Septic; Endotoxemia

INTERVENTIONS:
Device: TORAYMYXIN PMX-20R — Two (2) PMX cartridges will be administered approximately 24 hours apart. PMX Cartridge is an extracorporeal hemoperfusion device. Each treatment will target 2 hours with a minimum of 1 ½ hours, at a flow rate of approximately 100 ml/minute, (range of 80 to 120 ml/minute).

SUMMARY:
Open-label, non-controlled study of standard care plus the TORAYMYXIN PMX-20R (PMX cartridge) in subjects who have endotoxemia and septic shock. This is a continued access study subsequent to the EUPHRATES clinical trial NCT01046669.

DETAILED DESCRIPTION:
This is an open-label, non-controlled trial of standard medical care plus the TORAYMYXIN PMX-20R (PMX cartridge), in subjects with endotoxemia and septic shock. Subjects in ICUs will be assessed for septic shock using known or suspected infection and hypotension requiring vasopressor support as primary criteria. Endotoxemia will be assessed using the Endotoxin Activity Assay. Consented eligible subjects will receive two interventions with the PMX cartridge approximately 24 hours apart.The status of all subjects will be followed for 28 days, and long term follow-ups completed at 3 months, 6 months and 12 months.

This is a continued access study subsequent to the EUPHRATES clinical trial NCT01046669.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet the following criteria (and have a signed informed consent) will be allowed into the study:

1. Age ≥18 years of age
2. Hypotension requiring vasopressor support: Requirement for at least one of the vasopressors listed below, at the dose shown below, for at least 2 continuous hours and no more than 30 hours

   1. Norepinephrine > 0.05mcg/kg/min
   2. Dopamine > 10 mcg/kg/min
   3. Phenylephrine > 0.4 mcg/kg/min
   4. Epinephrine > 0.05 mcg/kg/min
   5. Vasopressin > 0.03 units/min
   6. Vasopressin (any dose) in combination with another vasopressor listed above
3. The subject must have received intravenous fluid resuscitation of a minimum of 30mL/kg administered within 24 hours of eligibility
4. Documented or suspected infection defined as definitive or empiric intravenous antibiotic administration
5. Endotoxin Activity Assay ≥ 0.60 EAA units
6. Evidence of at least 1 of the following criteria for new onset organ dysfunction that is considered to be due to the acute illness

   1. Requirement for positive pressure ventilation via an endotracheal tube or tracheostomy tube
   2. Thrombocytopenia defined as acute onset of platelet count < 150,000 μ/L or a reduction of 50% from prior known levels
   3. Acute oliguria defined as urine output < 0.5 ml/kg/hr for at least 6 hours despite adequate fluid resuscitation

Exclusion Criteria:

1. Inability to obtain an informed consent from the subject, family member or an authorized surrogate
2. Lack of commitment for full medical support
3. Inability to achieve or maintain a minimum mean arterial pressure (MAP) of ≥ 65mmHg despite vasopressor therapy and fluid resuscitation
4. Subject has end-stage renal disease and requires chronic dialysis
5. There is clinical support for non-septic shock such as:

   1. Acute pulmonary embolus
   2. Transfusion reaction
   3. Severe congestive heart failure (e.g. NYHA Class IV, ejection fraction < 35%)
6. Subject has had chest compressions as part of CPR during this hospitalization without immediate return to communicative state
7. Subject has had an acute myocardial infarction (AMI) within the past 4 weeks
8. Subject has uncontrolled hemorrhage (acute blood loss requiring > 3 UPC in the past 24 hours)
9. Major trauma within 36 hours of screening
10. Subject has severe granulocytopenia (leukocyte count less than 500 cells/mm3) or severe thrombocytopenia (platelet count less than 30,000 cells/mm3)
11. HIV infection in association with a last known or suspected CD4 count of <50/mm3
12. Subject's baseline state is non-communicative
13. Subject has sustained extensive third-degree burns within the past 7 days
14. Body weight < 35 kg (77 pounds)
15. Known hypersensitivity to Polymyxin B
16. Subject has known sensitivity or allergy to heparin or has a history of heparin associated thrombocytopenia (H.I.T.)
17. Subject is currently enrolled in an investigational drug or device trial
18. Subject has been previously enrolled in the current trial
19. Any other condition, that in the opinion of the investigator, would preclude the subject from being a suitable candidate for enrollment, such as end-stage chronic illness with no reasonable expectation of survival to hospital discharge
20. Subject has a screening MOD score ≤9

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult